CLINICAL TRIAL: NCT00233779
Title: Sirolimus-Eluting, Heparin-Coated Cobalt Chromium Balloon-Expandable Stent in the Treatment of Patients With de Novo Coronary Artery Lesions in Small Vessels (EVOLUTION)
Brief Title: Evaluation of Sirolimus-Eluting, Heparin-Coated CoCr Stent in the Treatment of de Novo Coronary Artery Lesions in Small Vessels(EVOLUTION)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P03-7401
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2007-06-27 (Estimated); Status verified 2007-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: SIROLIMUS-ELUTING, HEPARIN-COATED CoCr BALLOON-EXPANDABLE STENT

SUMMARY:
The objective of this study is to assess the performance and safety of a sirolimus-eluting, heparin-coated, cobalt chromium balloon-expandable stent (Small Vessel Stent) in patients with de novo native coronary artery lesions in small vessels as compared to historical data from small vessel patients in the RAVEL trial receiving the Sirolimus-eluting Bx VELOCITY™ stent.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be minimum 18 years of age;
2. Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II-III) OR patients with documented silent ischemia;

3 Treatment of one lesion in a native coronary artery. The treated lesion will be the one with the highest % diameter stenosis by visual estimate. Additional study stents may be used for procedural complications such as dissections. Multivessel treatment is permissible in non-target vessels; however, additional lesions may only be treated with commercial stents. If other non-target vessels are treated with commercial stents during the index procedure, they must be successfully treated prior to the study lesion;

4. The target lesion is >/=2.0 mm and </=2.5mm in diameter (visual estimate);

5. The target lesion can be covered with a single 18mm stent;

6. Target lesion stenosis is >50% and <100% (TIMI I) (visual estimate);

Exclusion Criteria:

1. Patient has experienced a Q-wave or non-Q-wave myocardial infarction with documented total CK>2 times normal within the preceding 24 hours and the CK and CK-MB enzymes remain above normal at the time of treatment;
2. Target lesion is due to in-stent restenosis;
3. Ejection fraction 30%;
4. Totally occluded vessel (TIMI 0 level);
5. Impaired renal function (creatinine > 3.0 mg/dL);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-10; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is in-stent late loss as measured by quantitative coronary angiography (QCA) at 6 months post-procedure. | 6 months post-procedure

SECONDARY OUTCOMES:
In-lesion late loss as measured by QCA at 6 months post-procedure. | 6 months post-procedure
In-stent and in-lesion minimum lumen diameter (MLD) and percent diameter stenosis (%DS) by QCA post-procedure and at 6 months. | Post-procedure and at 6 months
Device success defined as achievement of a final residual diameter stenosis of <50% (by QCA), using the assigned device only. If QCA is not available, the visual estimate of diameter stenosis is used.
Target Lesion Revascularization (TLR) at six and 12 months. | 6 and 12 months
Target Vessel Revascularization (TVR) at six and 12 months. | 6 and 12 months
Composite of Major Adverse Cardiac Events (MACE) defined as death, myocardial infarction (Q wave and non-Q wave), emergent bypass surgery, or repeat target lesion revascularization at 30 days, 6 months and 12 months post-procedure. | 30 days, 6 months and 12 months post-procedure
Stent Lumen and Stent Obstruction Volume by Intravascular Ultrasound (IVUS) at post procedure and six months follow-up. | post procedure and six months

CONTACTS AND LOCATIONS:
Overall Officials: J. E. Sousa, MD, Principal Investigator — Instituto Dante Pazzanese de Cardiologia
Locations (1):
- Instituto Dante Pazzanese de Cardiologia, São Paulo, Brazil